CLINICAL TRIAL: NCT05259917
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3, Three-way Crossover Trial to Evaluate the Efficacy and Safety of Two Dose Levels of KVD900, an Oral Plasma Kallikrein Inhibitor, for On-Demand Treatment of Angioedema Attacks in Adolescent and Adult Patients With Hereditary Angioedema Type I or II
Brief Title: A Phase III, Crossover Trial Evaluating the Efficacy and Safety of KVD900 (Sebetralstat) for On-Demand Treatment of Angioedema Attacks in Adolescent and Adult Patients With Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KVD900-301
Record Dates: First submitted 2022-02-04; First posted 2022-03-02 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Angioedema
Keywords: KONFIDENT; Sebetralstat
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KVD900 600 mg (Experimental)
  Interventions: Drug: KVD900 600 mg
- KVD900 300 mg (Experimental)
  Interventions: Drug: KVD900 300 mg

INTERVENTIONS:
Drug: Placebo — Placebo to KVD900 Tablet
  Arms: Placebo
Drug: KVD900 600 mg — KVD900 Tablet 600 mg (2 x 300 mg)
  Arms: KVD900 600 mg
Drug: KVD900 300 mg — KVD900 Tablet 300 mg (1 x 300 mg)
  Arms: KVD900 300 mg

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, phase III, three-way crossover clinical trial evaluating the efficacy and safety of KVD900, in the treatment of hereditary angioedema attacks in adolescent and adult Patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 12 years of age and older.
* Confirmed diagnosis of HAE type I or II at any time in the medical history.
* Patient has access to and ability to use conventional on-demand treatment for HAE attacks.
* If a patient is receiving long-term prophylactic treatment with one of the protocol-allowed therapies, they must be on a stable dose and regimen for at least 3 months prior to the Screening Visit (except for danazol, which requires a stable dose and regimen for 6 months prior to the Screening Visit). Patient must be willing to remain on a stable dose and regimen for the duration of the trial.
* Patient's last dose of attenuated androgens other than danazol was at least 28 days prior to randomization.
* Patient:

  1. has had at least 2 documented HAE attacks within 3 months prior to screening or randomization; or
  2. is a completer of the KVD824-201 trial within 3 months prior to randomization and meets all other entry criteria to enroll in KVD900-301
* Patients must meet the contraception requirements.
* Patients must be able to swallow trial tablets whole.
* Patients, as assessed by the Investigator, must be able to appropriately receive and store IMP, and be able to read, understand, and complete the electronic diary (eDiary).
* Investigator believes that the patient is willing and able to adhere to all protocol requirements.
* Patient provides signed informed consent or assent (when applicable). A parent or legally authorized representative (LAR) must also provide signed informed consent when required.

Exclusion Criteria:

* Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1-inhibitor deficiency, HAE with normal C1-INH (previously known as HAE type III), idiopathic angioedema, or angioedema associated with urticaria.
* A clinically significant history of poor response to bradykinin receptor 2 (BR2) blocker, C1-INH therapy or plasma kallikrein inhibitor therapy for the management of HAE, in the opinion of the Investigator.
* Use of angiotensin-converting enzyme (ACE) inhibitors after the Screening Visit or within 7 days prior to randomization.
* Any estrogen containing medications with systemic absorption (such as oral contraceptives including ethinylestradiol or hormonal replacement therapy) within 7 days prior to the Screening Visit.
* Patients who require sustained use of strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers.
* Inadequate organ function, including but not limited to:

  1. Alanine aminotransferase (ALT) >2x upper limit of normal (ULN)
  2. Aspartate aminotransferase (AST) >2x ULN
  3. Bilirubin direct >1.25x ULN
  4. International normalized ratio (INR) >1.2
  5. Clinically significant hepatic impairment defined as a Child-Pugh B or C
* Any clinically significant comorbidity or systemic dysfunction, which in the opinion of the Investigator, would jeopardize the safety of the patient by participating in the trial.
* History of substance abuse or dependence that would interfere with the completion of the trial, as determined by the Investigator.
* Known hypersensitivity to KVD900 or placebo or to any of the excipients.
* Prior participation in trial KVD900-201.
* Participation in any gene therapy treatment or trial for HAE.
* Participation in any interventional investigational clinical trial (with the exception of KVD824-201), including an investigational COVID-19 vaccine trial, within 4 weeks of the last dosing of investigational drug prior to screening.
* Any pregnant or breastfeeding patient.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals, Ltd.
Locations (63):
- United States (21):
  - KalVista Investigative Site, Birmingham, Alabama
  - KalVista Investigative Site, Scottsdale, Arizona
  - KalVista Investigative Site, Little Rock, Arkansas
  - KalVista Investigative Site, San Diego, California
  - KalVista Investigative Site, Santa Monica, California
  - KalVista Investigative Site, Centennial, Colorado
  - KalVista Investigative Site, Colorado Springs, Colorado
  - KalVista Investigative Site, Tampa, Florida
  - KalVista Investigative Site, Chicago, Illinois
  - KalVista Investigative Site, Overland Park, Kansas
  - KalVista Investigative Site, Louisville, Kentucky
  - KalVista Investigative Site, Chevy Chase, Maryland
  - KalVista Investigative Site, Plymouth, Minnesota
  - KalVista Investigative Site, St Louis, Missouri
  - KalVista Investigative Site, New York, New York
  - KalVista Investigative Site, Charlotte, North Carolina
  - KalVista Investigative Site, Toledo, Ohio
  - KalVista Investigative Site, Hershey, Pennsylvania
  - KalVista Investigative Site, Dallas, Texas
  - KalVista Investigative Site, Layton, Utah
  - KalVista Investigative Site, Spokane, Washington
- KalVista Investigative Site, Campbelltown, New South Wales, Australia
- KalVista Investigative Site, Sofia, Bulgaria
- KalVista Investigative Site, Toronto, Ontario, Canada
- France (3):
  - KalVista Investigative Site, Grenoble
  - KalVista Investigative Site, Lille
  - KalVista Investigative Site, Paris
- Germany (4):
  - KalVista Investigative Site, Frankfurt am Main, Hesse
  - KalVista Investigative Site, Berlin
  - KalVista Investigative Site, Mainz
  - KalVista Investigative Site, Mörfelden-Walldorf
- Greece (2):
  - Kalvista Investigative Site, Athens
  - KalVista Investigative Site, Athens
- KalVista Investigative Site, Budapest, Hungary
- Israel (4):
  - KalVista Investigative Site, Haifa
  - KalVista Investigative Site, Petach Tikvah
  - KalVista Investigative Site, Ramat Gan
  - KalVista Investigative Site, Tel Aviv
- Italy (2):
  - KalVista Investigative Site, Padua
  - KalVista Investigative Site, San Donato Milanese
- Japan (6):
  - KalVista Investgative Site, Takatsuki-shi, Osaka
  - KalVista Investgative Site, Chiba
  - KalVista Investigative Site, Gunma
  - KalVista Investigative Site, Hiroshima
  - KalVista Investigative Site, Saitama
  - KalVista Investigative Site, Yokohama
- KalVista Investigative Site, Amsterdam, Netherlands
- KalVista Investigative Site, Auckland, New Zealand
- KalVista Investigative Site, Skopje, North Macedonia
- Poland (3):
  - KalVista Investigative Site, Bialystok
  - KalVista Investigative Site, Krakow
  - KalVista Investigative Site, Lodz
- KalVista Investigative Site, Porto, Portugal
- KalVista Investigative Site, San Juan, Puerto Rico
- KalVista Investigative Site, Sângeorgiu de Mureş, Mureș County, Romania
- KalVista Investigative Site, Martin, Slovakia
- Spain (2):
  - KalVista Investigative Site, Barcelona
  - KalVista Investigative Site, Madrid
- United Kingdom (5):
  - KalVista Investigative Site, Birmingham
  - KalVista Investigative Site, Cardiff
  - KalVista Investigative Site, Frimley
  - KalVista Investigative Site, Leeds
  - KalVista Investigative Site, London

IPD SHARING:
Plan to Share IPD: No
Data will not be shared until all global regulatory filings are complete

REFERENCES:
- [Background] Riedl MA, Farkas H, Aygoren-Pursun E, Psarros F, Soteres DF, Staevska M, Cancian M, Hagin D, Honda D, Melamed I, Savic S, Stobiecki M, Busse PJ, Dias de Castro E, Agmon-Levin N, Gower R, Kessel A, Kurowski M, Lleonart R, Grivcheva Panovska V, Wedner HJ, Audhya PK, Hao J, Iverson M, Smith MD, Yea CM, Lumry WR, Zanichelli A, Bernstein JA, Maurer M, Cohn DM; KONFIDENT Investigators. Oral Sebetralstat for On-Demand Treatment of Hereditary Angioedema Attacks. N Engl J Med. 2024 Jul 4;391(1):32-43. doi: 10.1056/NEJMoa2314192. Epub 2024 May 31. PMID 38819658
- [Derived] Farkas H, Anderson J, Bouillet L, Caballero T, Cancian M, Craig T, Fukunaga A, Grivcheva-Panovska V, Guilarte M, Honda D, Kanarek H, Kiani-Alikhan S, Kinaciyan T, Leguevaques D, Longhurst HJ, Magerl M, Manning ME, Martinez-Saguer I, Melamed I, O'Connor ME, Peter J, Savic S, Soteres DF, Staevska M, Staubach P, Stobiecki M, Tachdjian R, Valerieva A, Yong PFK, Hao J, Iverson M, Smith MD, Yea CM, Audhya PK, Aygoren-Pursun E, Bernstein JA, Cohn DM, Lumry WR, Riedl MA, Zanichelli A, Maurer M. Long-Term Safety and Effectiveness of Sebetralstat: Interim Analysis of KONFIDENT-S Open-label Extension. J Allergy Clin Immunol Pract. 2025 Nov;13(11):3094-3103.e5. doi: 10.1016/j.jaip.2025.08.020. Epub 2025 Aug 29. PMID 40886933
- [Derived] Aygoren-Pursun E, Zanichelli A, Cohn DM, Cancian M, Hakl R, Kinaciyan T, Magerl M, Martinez-Saguer I, Stobiecki M, Farkas H, Kiani-Alikhan S, Grivcheva-Panovska V, Bernstein JA, Li HH, Longhurst HJ, Audhya PK, Smith MD, Yea CM, Maetzel A, Lee DK, Feener EP, Gower R, Lumry WR, Banerji A, Riedl MA, Maurer M. An investigational oral plasma kallikrein inhibitor for on-demand treatment of hereditary angioedema: a two-part, randomised, double-blind, placebo-controlled, crossover phase 2 trial. Lancet. 2023 Feb 11;401(10375):458-469. doi: 10.1016/S0140-6736(22)02406-0. PMID 36774155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 158 patients were screened, of which 22 were screen failures. The majority of screen failures were due to inclusion criterion not met.
Pre-assignment Details: A total of 136 patients were randomized across the 6 treatment sequences in a 3-way crossover design, of which a total of 110 patients treated at least 1 attack with IMP and therefore were included in the Full Analysis Set (FAS).
Groups:
- Sequence A: PLB/600 mg KVD900/300 mg KVD900
- Sequence B: PLB/ 300 mg KVD900/ 600 mg KVD900
- Sequence C: 300 mg KVD900/ 600 mg KVD900/PLB
- Sequence D: 300 mg KVD900/PLB/ 600 mg KVD900
- Sequence E: 600 mg KVD900/ 300 mg KVD900/PLB
- Sequence F: 600 mg KVD900/PLB/ 300 mg KVD900
Period: Overall Study
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 18 | 18 | 15 | 17 | 20 | 22
Completed (Completed - defined as treating 3 attacks with IMP. Trial Termination by Sponsor, defined as ongoing patients terminated once the trial objectives were met.) | 10 | 14 | 8 | 12 | 8 | 16
Not Completed | 8 | 4 | 7 | 5 | 12 | 6
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Trial Termination by Sponsor | 7 | 2 | 3 | 5 | 11 | 4
Not completed — Other | 1 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F | Total
Number analyzed (Participants) | 18 | 18 | 15 | 17 | 20 | 22 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (15.70) | 35.8 (16.90) | 41.1 (17.87) | 31.8 (11.42) | 41.4 (14.60) | 38.2 (13.14) | 37.7 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 5 | 12 | 11 | 11 | 66
  Male | 5 | 4 | 10 | 5 | 9 | 11 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 1 | 2 | 0 | 7
  Not Hispanic or Latino | 15 | 17 | 10 | 15 | 17 | 21 | 95
  Unknown or Not Reported | 2 | 1 | 2 | 1 | 1 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 5 | 1 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 14 | 18 | 12 | 11 | 18 | 19 | 92
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 1 | 2 | 7
Height [Mean (Standard Deviation); unit: meters] | 1.646 (0.1216) | 1.694 (0.1135) | 1.715 (0.0877) | 1.657 (0.1205) | 1.686 (0.0884) | 1.704 (0.1126) | 1.684 (0.1088)
Weight [Mean (Standard Deviation); unit: kilograms] | 75.16 (16.109) | 73.88 (16.603) | 83.80 (18.157) | 72.28 (23.735) | 77.90 (16.321) | 83.55 (21.949) | 77.86 (19.179)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.78 (5.638) | 25.62 (4.743) | 28.62 (6.603) | 26.15 (7.701) | 27.37 (5.162) | 28.90 (7.329) | 27.44 (6.261)
Treatment Regimen [Count of Participants; unit: Participants]
  Prophylaxis | 3 | 5 | 3 | 3 | 3 | 7 | 24
  On Demand Only | 15 | 13 | 12 | 14 | 17 | 15 | 86

OUTCOME MEASURES:

1. Primary Outcome: Time to Beginning of Symptom Relief Patient Global Impression of Change (PGI-C)
Description: The analysis of time to the beginning of symptom relief defined as at least "a little better" (2 time points in a row) on the PGI-C within 12 hours of the first IMP administration using the Gehan score transformation test for Full Analysis Set (FAS).
  Attacks were treated as right-censored at 12 hours if they did not achieve beginning of symptom relief defined by PGI-C as at least "a little better" (2 time points in a row) or received conventional attack treatment prior to time-to-event within 12 hours of the first IMP administration.
  When an endpoint result was non-evaluable (NE) within 12 hours, if the event did occur, the event must have occurred >12 hours following study drug.
Time Frame: Within 12 hours of the first investigational medicinal product (IMP) administration.
Population: The full analysis set (FAS) included all randomized patients who received trial medication from at least one period for the respective qualifying HAE attack and are presented according to the randomized treatment. The FAS was the population for efficacy analyses.
Measure: Median (95% Confidence Interval); unit: Time (h)
Groups:
- KVD900 600 mg: KVD900 600 mg: Two KVD900 Tablets 300 mg (2 x 300 mg)
Arm/Group | KVD900 300 mg | KVD900 600 mg | Placebo
Number analyzed (Participants) | 87 | 93 | 84
Time (h) | 1.61 [1.28 to 2.27] | 1.79 [1.33 to 2.27] | 6.72 [2.33 to NA] — NA represents non-evaluable (NE), defined as subjects not reaching at least "a little better" (2 time points in a row) on the PGI-C within 12 hours of the first IMP administration to complete descriptive statistics.
Statistical Analysis 1: Comparison: KVD900 300 mg vs Placebo; Gehan score transformation test: KVD900 300 mg vs Placebo; Test type: Superiority; p < 0.0001, Gehan score transformation test
Statistical Analysis 2: Comparison: KVD900 600 mg vs Placebo; Gehan score transformation test: KVD900 600 mg vs Placebo; Test type: Superiority; p = 0.0013, Gehan score transformation test

2. Secondary Outcome: Time to First Incidence of Decrease From Baseline Patient Global Impression of Severity (PGI-S) (2 Time Points in a Row)
Description: First incidence of decrease in attack severity at two time points in a row (with possible missing values in between) within 12 hours of the first IMP administration.
  Attacks were treated as right-censored at 12 hours if they did not have a decrease in PGI-S score from baseline for 2 time points in a row or received conventional attack treatment prior to time-to-event within 12 hours of the first IMP administration.
  When an endpoint result was non-evaluable (NE) within 12 hours, if the event did occur, the event must have occurred >12 hours following study drug.
Time Frame: Within 12 hours of the first IMP administration.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Time (h)
Arm/Group | KVD900 300 mg | KVD900 600 mg | Placebo
Number analyzed (Participants) | 87 | 93 | 84
Time (h) | 9.27 [4.08 to NA] — NA represents non-evaluable (NE), defined as subjects not reaching first incidence of decrease from baseline Patient Global Impression of Severity (PGI-S) within 12 hours of the first IMP administration to complete descriptive statistics. | 7.75 [3.27 to NA] — NA represents non-evaluable (NE), defined as subjects not reaching first incidence of decrease from baseline Patient Global Impression of Severity (PGI-S) within 12 hours of the first IMP administration to complete descriptive statistics. | NA [NA to NA] — NA represents non-evaluable (NE), defined as subjects not reaching first incidence of decrease from baseline Patient Global Impression of Severity (PGI-S) within 12 hours of the first IMP administration to complete descriptive statistics.
Statistical Analysis 1: Comparison: KVD900 300 mg vs Placebo; Gehan score transformation test: KVD900 300 mg vs Placebo; Test type: Superiority; p = 0.0036, Gehan score transformation test
Statistical Analysis 2: Comparison: KVD900 600 mg vs Placebo; Gehan score transformation test: KVD900 600 mg vs Placebo; Test type: Superiority; p = 0.0032, Gehan score transformation test

3. Secondary Outcome: Time to Complete HAE Attack Resolution (PGI-S)
Description: Time to complete HAE attack resolution defined as "none".
  Attacks were treated as right-censored at 24 hours if they did reach complete HAE attack resolution or received conventional attack treatment prior to time-to-event within 24 hours of IMP administration.
  When an endpoint result was non-evaluable (NE) within 24 hours, if the event did occur, the event must have occurred >24 hours following study drug.
Time Frame: Within 24 hours of the first IMP administration.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Time (h)
Arm/Group | KVD900 300 mg | KVD900 600 mg | Placebo
Number analyzed (Participants) | 87 | 93 | 84
Time (h) | NA [16.60 to NA] — NA represents non-evaluable (NE), defined as not reaching complete HAE attack resolution defined as "none" within 24 hours of the first IMP administration to complete descriptive statistics. | 24.00 [10.60 to NA] — NA represents non-evaluable (NE), defined as not reaching complete HAE attack resolution defined as "none" within 24 hours of the first IMP administration to complete descriptive statistics. | NA [NA to NA] — NA represents non-evaluable (NE), defined as not reaching complete HAE attack resolution defined as "none" within 24 hours of the first IMP administration to complete descriptive statistics.
Statistical Analysis 1: Comparison: KVD900 300 mg vs Placebo; Gehan score transformation test: KVD900 300 mg vs Placebo; Test type: Superiority; p = 0.0022, Gehan score transformation test
Statistical Analysis 2: Comparison: KVD900 600 mg vs Placebo; Gehan score transformation test: KVD900 600 mg vs Placebo; Test type: Superiority; p < 0.0001, Gehan score transformation test

ADVERSE EVENTS:
Time Frame: The period of observation for AEs extends from the time of the patient's first dose of IMP until the Final/ET Visit, an average of 18 weeks.
Description: Ongoing AEs at the Final/ET Visit will be followed up until the AE has resolved or is considered chronic or stable or the AE has been clearly shown to be unrelated to the IMP. The period of observation for SAEs extends from the time of signing the informed consent until the Final/ET Visit.
Arm/Group | KVD900 300 mg | KVD900 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/93 | 0/83
Serious Adverse Events (participants affected / at risk) | 1/86 | 2/93 | 0/83
Other Adverse Events (participants affected / at risk) | 5/86 | 6/93 | 13/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KVD900 300 mg (N=86) | KVD900 600 mg (N=93) | Placebo (N=83)
HEREDITARY ANGIOEDEMA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
ANISOCORIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KVD900 300 mg (N=86) | KVD900 600 mg (N=93) | Placebo (N=83)
EYE HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT05259917/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT05259917/SAP_001.pdf